CLINICAL TRIAL: NCT06812988
Title: A 52-week Randomized, Double-blind, Placebo-controlled, Multi-center Phase 2a Study Assessing Safety and Efficacy of SAR442970, a Dual Anti-TNF-α and Anti-OX40L NANOBODY® Molecule, for Preservation of Pancreatic β-cell Function in Adults and Adolescents With Recently Diagnosed Type 1 Diabetes
Brief Title: Treatment of Type 1 Diabetes With Anti-OX40L Bispecific With Anti-TNF Activity In a Single Nanobody® Molecule
Acronym: T1D OBTAIN
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACT18368; U1111-1307-7268 (Other: WHO ICTRP)
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SAR442970 (Experimental): Participants will receive subcutaneous injection of SAR442970.
  Interventions: Drug: SAR442970
- Placebo (Placebo Comparator): Participants will receive subcutaneous injection of matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAR442970 — Pharmaceutical form: Solution Route of administration: Subcutaneous injection
  Arms: SAR442970
Drug: Placebo — Pharmaceutical form: Solution Route of administration: Subcutaneous injection
  Arms: Placebo

SUMMARY:
This is a randomized, placebo-controlled, parallel group, multicenter, double-blind Phase 2a, 2-arm study.

The goal of this Phase 2a study is to assess safety and efficacy of SAR442970 in comparison to placebo to preserve β-cell function in participants with recently diagnosed type 1 diabetes (T1D) on insulin therapy.

The study design comprises 2 parts: in Part A adult participants (18 to 35 years of age at screening) and in Part B adolescent and young adult participants (age range 12 to 21 years) will be randomized into SAR442970 and placebo groups. Approximately 84 participants will be included with randomization ratio 3:1 (active:placebo).

The study includes a screening period (3 to 5 weeks), a double-blind treatment period of 52 weeks and a safety follow-up of 26 weeks.

DETAILED DESCRIPTION:
The total study duration will be up to 83 weeks including Screening and Safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 18 to 35 y.o. inclusive, at the time of signing the informed consent in order to be enrolled in Part A. Participant must be 12 to 21 y.o. inclusive, at the time of signing the informed consent in order to be enrolled in Part B.
2. Participants who meet the criteria of T1D according to American Diabetes Association (ADA 2024).
3. Initiated exogenous insulin replacement therapy not longer than 90 days prior to Screening visit at which random C-peptide will be assessed.
4. Receiving insulin hormone replacement therapy:
5. Participants must be positive for at least 1 of the following T1D autoantibodies confirmed by medical history and/or obtained at study Screening:

   * Glutamic acid decarboxylase (GAD-65)
   * Insulinoma Antigen-2 (IA-2)
   * Zinc-transporter 8 (ZnT8) or
   * Insulin (if obtained not later than 10 days after exogenous insulin therapy initiation)
6. Have random C-peptide levels ≥0.2 nmol/L determined at Screening.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Serious systemic viral, bacterial or fungal infection (eg, pneumonia, pyelonephritis), infection requiring hospitalization or intravenous (IV) antibiotics or significant chronic viral (including history of recurrent or active herpes zoster, acute or active cytomegalovirus [CMV], Epstein-Barr Virus [EBV] as determined at Screening), bacterial, or fungal infection (eg, osteomyelitis) 30 days before and during Screening.
2. History of invasive opportunistic infections, such as, but not limited to histoplasmosis, listeriosis, coccidioidomycosis, candidiasis, pneumocystis jirovecii, and aspergillosis, regardless of resolution.
3. Evidence of active or latent tuberculosis (TB) as documented by medical history and examination, chest X-rays (posterior anterior and lateral), and/or TB testing.
4. Evidence of any clinically significant, severe or unstable, acute or, chronically progressive, uncontrolled infection, medical or surgical condition (eg, but not limited to, cerebral, cardiac, pulmonary, renal, hepatic, gastrointestinal, neurologic, or any known immune deficiency), or any condition that may affect participant safety in the judgment of the Investigator (including vaccinations which are not updated based on local regulation).
5. History of a systemic hypersensitivity reaction or significant allergies, other than localized injection site reaction, to any humanized mAb. Clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe post-treatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear IgA dermatosis, toxic epidermal necrolysis, and exfoliative dermatitis).
6. History of moderate to severe congestive heart failure (New York Health Association [NYHA] Class III or IV), or recent cerebrovascular accident, or any other condition which, in the opinion of the Investigator, would put the participant at risk by participation in the protocol.
7. History of demyelinating disease (including myelitis) or neurologic symptoms suggestive of demyelinating disease.
8. Has other autoimmune or inflammatory conditions
9. Diabetes of forms other than autoimmune T1D that include but are not limited to genetic forms of diabetes, maturity-onset diabetes of the young (MODY), latent autoimmune diabetes of the adult (LADA), secondary to medications or surgery, type 2 diabetes by judgment of the investigator.
10. History of malignancy or lymphoproliferative disease other than adequately treated localized carcinoma in situ of the cervix or nonmetastatic squamous cell carcinoma, or nonmetastatic basal cell carcinoma of the skin that was excised and completely cured or any family history in two or more relatives (immediate family) of same cancer (ie, rare cancers, those manifesting at a young age in a parent or sibling, certain genetic-based inheritable cancers).
11. Systemic corticosteroids (duration >7 days), adrenocorticotropic hormone 1 month prior to Screening.
12. Any IV, intramuscular (IM) or SC administered biologic treatments (mono- or polyclonal antibodies affecting function of immune system), <3 months or <5 half-lives (whichever is longer), prior to randomization.
13. Any live (attenuated or viral-vector) vaccine (including but not limited to varicella zoster, oral polio, nasal influenza, rabies) within 3 months prior to randomization or is scheduled in expected period of study (78 weeks after randomization) if this vaccination cannot be safely postponed.
14. Any non-live (inactivated, mRNA, recombinant, conjugate, toxoid) vaccine administered less than 14 days prior to randomization.
15. Any immunosuppressive therapy within 12 weeks prior to randomization and through 78 weeks after randomization
16. Course of Thymoglobulin®, teplizumab or other immunomodulatory treatments at any time
17. Any drugs that may be used for treatment of T1D and type 2 diabetes other than insulin including but not limited to metformin, glucagon-like peptide 1 (GLP-1) agonists, sodium-glucose co-transporter-2 and 1 (SGLT2/1) inhibitor, and verapamil within 2 weeks prior to Screening.
18. Abnormal laboratory test(s) at Screening
19. Participants who have impaired renal function with estimated glomerular filtration rate (eGFR) (using the Modification of Diet in Renal Disease [MDRD] formula) <60 mL/min/1.73 m2, or using the bedside Schwartz equation in the participants under the age of 18 y.o.

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2027-04-29 (Estimated); Study Completion 2027-04-29 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to Week 26 in mean 2-hour mixed meal tolerance test (MMTT) stimulated C-peptide concentration | From Baseline to Week 26
  Mixed meal tolerance test MMTT stimulated C-peptide concentration is to be calculated from area under the concentration-time curve (AUC)

SECONDARY OUTCOMES:
Change from baseline to Week 52 in mean 2-hour MMTT stimulated Cpeptide concentration | From Baseline to Week 52
  MMTT stimulated C-peptide concentration is to be calculated from area under the concentration-time curve (AUC)
Participant remaining C-peptide positive at Week 26 and Week 52 | Week 26 and Week 52
  Incidence (yes/no) outcome Defined as mean 2-hour MMTT stimulated C-peptide concentration ≥0.2 nmol/L
Time in range (TIR) (70-180 mg/dL) at Week 26 and Week 52 | Week 26 and Week 52
  Assessed by Continuous glucose monitoring (CGM). A CGM system is a device that records interstitial glucose levels continuously throughout the day and night via a subcutaneous sensor.
Change from baseline to Week 26 and Week 52 in insulin dose | From Baseline to Week 26 and Week 52
  Expressed in IU/kg/day
Change from baseline to Week 26 and Week 52 in glycated hemoglobin A1c (HbA1c) level | From Baseline to Week 26 and Week 52
Participant having HbA1c ≤6.5% and ≤0.25 IU/kg/day of exogenous insulin required at Week 26 and Week 52 | Week 26 and Week 52
  Incidence (yes/no) outcome
Incidence of treatment emergent adverse events (TEAEs), serious adverse events (SAEs), adverse events of special interest (AESIs) and TEAEs leading to treatment discontinuation | Up to End of Study (approx. 83 Weeks)
Incidence (yes/no) of hypoglycemic events (level 2 or 3 according to American Diabetes Association) | Up to End of Study (approx. 83 Weeks)
  Incidence (yes/no) outcome
Incidence (yes/no) of hyperglycemic episodes (level 2 according to American Diabetes Association) | Up to End of Study (approx. 83 Weeks)
  Incidence (yes/no) outcome
Incidence (yes/no) of diabetic ketoacidosis (DKA) events | Up to End of Study (approx. 83 Weeks)
  Incidence (yes/no) outcome
Incidence (yes/no) of clinically significant changes in vital signs, electrocardiogram (ECG), and/or laboratory evaluation | Up to End of Study (approx. 83 Weeks)
  Incidence (yes/no) outcome
SAR442970 serum concentrations over time | Up to End of Study (approx. 83 Weeks)
Incidence of anti-drug antibodies (ADAs) over time | Up to End of Study (approx. 83 Weeks)
Change from baseline to Week 26 and Week 52 in Problem Areas in Diabetes (PAID) total score (all participants) | From Baseline to Week 26 and Week 52
  The Problem Areas in Diabetes (PAID) is a diabetes specific instrument measuring diabetes distress. There is an adult version (18+) and a pediatric version for children 8-17 years of age. The PAID contains 20 items that describe negative emotions related to diabetes (eg, depression, anger, frustration). Item scores are summed to generate a total score. Scores range from 0 to 100, where higher total scores correspond to higher emotional distress due to diabetes
Change from baseline to Week 26 and Week 52 in PAID immediate and theoretical domain scores (caregivers of all participants 12 to 17 y.o.) | From Baseline to Week 26 and Week 52
  Caregiver version of PAID for parents with children 8-18 years of age consists of 18 items that measure caregiver burden. Two scores are calculated: Immediate Burden and Theoretical Burden. Scores range from 0 to 100, where higher scores correspond to greater caregiver burden.

CONTACTS AND LOCATIONS:
Locations (24):
- United States (5):
  - Atlanta Diabetes Associates- Site Number : 8400006, Atlanta, Georgia
  - IACT Health - Columbus - Talbotton Road- Site Number : 8400012, Columbus, Georgia
  - Profound Research - MHP - TriAtria- Site Number : 8400015, Farmington Hills, Michigan
  - Tekton Research - McKinney- Site Number : 8400017, McKinney, Texas
  - Advanced Research Institute - Odgen- Site Number : 8400007, Ogden, Utah
- Argentina (5):
  - Investigational Site Number : 0320001, Buenos Aires
  - Investigational Site Number : 0320002, Buenos Aires
  - Investigational Site Number : 0320005, Buenos Aires
  - Investigational Site Number : 0320004, Buenos Aires
  - Investigational Site Number : 0320003, Salta
- Australia (3):
  - Investigational Site Number : 0360003, Saint Leonards, New South Wales
  - Investigational Site Number : 0360002, Brisbane, Queensland
  - Investigational Site Number : 0360001, Parkville, Victoria
- Brazil (2):
  - Centro de Diabetes Curitiba- Site Number : 0760005, Curitiba, Paraná
  - Centro de Pesquisas Clínicas - São Paulo- Site Number : 0760002, São Paulo
- Canada (2):
  - Investigational Site Number : 1240006, Surrey, British Columbia
  - Investigational Site Number : 1240001, Vancouver, British Columbia
- Chile (3):
  - Investigational Site Number : 1520003, Providencia, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520004, Concepción, Región del Biobío
- Israel (3):
  - Investigational Site Number : 3760001, Jerusalem
  - Investigational Site Number : 3760003, Kefar Sava
  - Investigational Site Number : 3760002, Ramat Gan
- Investigational Site Number : 6820002, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: ACT18368 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26518&tenant=MT_SNY_9011